CLINICAL TRIAL: NCT06144554
Title: Post Market Registry to Collect Real-World Safety and Effectiveness Data for the Omnipod 5 System in Children and Adults With Type 1 Diabetes
Brief Title: Post Market Registry for the Omnipod 5 System in Children and Adults With Type 1 Diabetes
Status: Recruiting | Type: Observational
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Post-Market Registry
Record Dates: First submitted 2023-11-10; First posted 2023-11-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Omnipod; Automated Insulin Delivery; Registry
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Omnipod User: All new users for the Omnipod 5 System will be required to register with Insulet's Podder Central. Users already in Podder Central will be required to log into their account before logging into the Omnipod 5 Controller if transitioning to the Omnipod 5 System. As part of the onboarding process, users will be invited to participate in this registry.
  Interventions: Device: Omnipod 5

INTERVENTIONS:
Device: Omnipod 5 — The Omnipod 5 System consists of a tubeless insulin Pod and the Omnipod® 5 App, installed on a designated Controller or compatible Android smartphone. The Omnipod 5 System works with the Dexcom G6® Continuous Glucose Monitoring System to continuously adapt and automatically deliver insulin according to personal needs.
  Every two weeks while on the Omnipod 5 system, participants will receive a push notification to complete assessments including any severe hypoglycemia or diabetic ketoacidosis events experienced since the prior assessment.

SUMMARY:
This is a decentralized observational clinical registry to collect real-world evidence related to the safety and effectiveness of the Omnipod 5 system in children and adults with Type 1 Diabetes.

DETAILED DESCRIPTION:
This is a decentralized observational clinical registry to collect real-world evidence related to the safety and effectiveness of the Omnipod 5 system in children and adults with Type 1 Diabetes.

A minimum of 2,200 Type 1 participants will be recruited to ensure a minimum of 1,650 participants completing 12 months of follow-up. The minimum number of completed participants is as follows:

* 150 participants aged 2-5
* 300 participants aged 6-13
* 300 participants aged 14-17
* 900 participants aged 18+

In addition to the enrollment targets above, a minimum of 1100 Omnipod-naïve users, 880 pump-naïve users, and 110 CGM-naïve users will be recruited.

Participants are expected to be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported type 1 diabetes
2. Prescribed, obtained, and have been using the Omnipod 5 System for no more than two weeks or plan to start using the system within the next two weeks
3. Willing to use only the following types of U-100 insulin during the study: Humalog U-100, Novolog, or Admelog
4. Able to read and speak English or Spanish (when available) fluently and reside full time in the United States
5. Willing to collect A1C samples using a provided home kit and send the samples to the registry specific core laboratory at baseline and 3, 6, 9 and 12 months
6. Willing and able to complete registry assessments every two weeks
7. Willing and able to complete registry outcome questionnaires at baseline, 6 months and end of study (or at withdrawal)
8. Is not currently pregnant or planning to become pregnant in the next 12 months and is using a reliable form of birth control
9. Access to internet via phone, tablet and/or computer to use the registry online platform
10. Willing to provide CGM and insulin delivery data collected prior to using the Omnipod 5 System, if available (participants will not be excluded if data is not provided)
11. Willing and able to provide informed consent (or assent) and/or has a parent/guardian willing and able to provide informed consent as applicable

Exclusion Criteria:

1. Diagnosed with sickle cell anemia and/or hemoglobinopathy
2. Planned blood transfusions over the course of the study or has received a blood transfusion within 3 months prior to starting on Omnipod 5
3. Adults that are unable to provide informed consent

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All new users for the Omnipod 5 System will be required to register with Insulet's Podder Central. Users already in Podder Central will be required to log into their account before logging into the Omnipod 5 Controller if transitioning to the Omnipod 5 System.
  A minimum of 2,200 Type 1 participants will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of severe hypoglycemia | From baseline to study completion, up to 12 months.
  Measures frequency of severe hypoglycemia
Incidence rate of DKA | From baseline to study completion, up to 12 months.
  Measures frequency of DKA
A1c at 3, 6, 9 and 12 months | Comparing the change in A1c at baseline compared to at 3, 6, 9 and 12 months
  Measures device effectiveness
Percentage of time < 54 mg/dL | From baseline to study completion, up to 12 months
  Glucose metric from study continuous glucose monitoring system
Percentage of time < 70 mg/dL | From baseline to study completion, up to 12 months
  Glucose metric from study continuous glucose monitoring system
Percentage of time > 180 mg/dL | From baseline to study completion, up to 12 months
  Glucose metric from study continuous glucose monitoring system
Percentage of time > 250 mg/dL | From baseline to study completion, up to 12 months
  Glucose metric from study continuous glucose monitoring system
Percentage of time in range 70-180 mg/dL | From baseline to study completion, up to 12 months
  Glucose metric from study continuous glucose monitoring system
Mean Glucose mg/dL | From baseline to study completion, up to 12 months
  Glucose metric from study continuous glucose monitoring system
Standard deviation of glucose mg/dL | From baseline to study completion, about 12 months
  measure of the range of glucose readings
Glucose management indicator % | From baseline to study completion, up to 12 months
  MI tells you what your approximate A1C level is likely to be, based on the average glucose level from your CGM readings for 14 or more days.
Percentage of participants achieving A1C < 7% | From baseline to study completion, up to 12 months
  measurement of percentage of participants with A1c less than 7%
Percentage of participants with time in range > 70% | From baseline to study completion, up to12 months
  measurement of percentage of participants with time in range > 70%
Percentage of participants with time below range (<70mg/dL) of < 4% | From baseline to study completion, up to 12 months
  measurement of percentage of participants with time below range (<70mg/dL) of < 4%
Insulin Usage | From baseline to study completion, up to 12 months
  Measure of insulin requirements
Body Mass Index (BMI) or BMI z-score | at 6 months and at the end of registry participation, up to 12 months.
  Changes in body mass index
EQ-5D (inclusive of the Visual Analogue Scale (VAS)) | at baseline, at 6 months and at the end of registry participation, up to 12 months.
  Questionaire
Insulin Delivery Systems: Perceptions, Ideas, Reflections, and Expectations (INSPIRE) | at baseline, at 6 months and at the end of registry participation, up to 12 months
  Questionaire
System Usability Scale (SUS) | at baseline, at 6 months and at the end of registry participation, up to 12 months
  Questionnaire
Incidence rate of prolonged hyperglycemia (events per person months) during usage of Activity Feature | From baseline to study completion, up to 12 months
  Measuring rate of prolonged high sugar while in activity feature
Incidence rate of prolonged hyperglycemia (events per person months) | From baseline to study completion, up to 12 months
  Measuring the occurrence of prolonged hyperglycemia
Incidence rate of prolonged hyperglycemia (events per person months) during usage of a Target Glucose of 140 mg/dL or 150 mg/dL | From baseline to study completion, up to 12 months
  Measuring the occurrence of prolonged hyperglycemia while at a set target glucose of 140mg/dL or 150mg/dL
Glucose Outcomes during the 4-hour post-bolus period using the SmartBolus Calculator: o Percentage of time < 54 mg/dL o Percentage of time in range 70-180 mg/dL | From baseline to study completion, up to 12 months
  Glucose metric from study CGM

CONTACTS AND LOCATIONS:
Locations (1):
- Circuit Clinical, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No